CLINICAL TRIAL: NCT06673407
Title: Pilot Trial on the Contribution of Peer Leaders and Self-Compassion to Group Exposure Workshops for Socially Anxious Undergraduates
Brief Title: Group Exposure Workshops for Socially Anxious Undergraduates
Acronym: OASIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Joanna Arch, Yvonne Kristy Endowed Chair, Renée Crown Wellness Institute; Professor, Department of Psychology and Neuroscience, University of Colorado, Boulder
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0178
Record Dates: First submitted 2024-10-08; First posted 2024-11-04 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Social Anxiety Disorder; Public Speaking Fear; Public Speaking Anxiety; Social Fear
Keywords: Social Anxiety; Public Speaking Anxiety; Exposure Therapy; Peer-led; Self-compassion; Common Humanity
MeSH Terms: conditions — Phobia, Social; Glossophobia

STUDY DESIGN:
Intervention Model Description: This trial uses a 2-variable full factorial design within the Multiphase Optimization Strategy (MOST) framework. Participants will be assigned to one of four study conditions involving 5.5-7.5-hours of workshops (depending on study condition) conducted over 3 in-person group sessions. Study conditions will vary depending on whether they 1) include self-compassion (i.e., common humanity) enhancements, and 2) are led by peer co-facilitators.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Exposure Only (Active Comparator): Group exposure therapy for social anxiety and public speaking fears.
  Interventions: Behavioral: Group Exposure for Social Anxiety
- Compassion Enhanced (Experimental): Group exposure therapy for social anxiety and public speaking fears plus self-compassion exercises aimed at inducing a sense of common humanity.
  Interventions: Behavioral: Self-Compassion Enhanced Group Exposure Therapy for Social Anxiety
- Peer enhanced (Experimental): Group exposure therapy for social anxiety and public speaking fears facilitated by a pair of doctoral student and undergraduate student co-facilitators who will explicitly use appropriate self-disclosure to establish the co-facilitators as individuals with lived experiences of social anxiety and public speaking fears.
  Interventions: Behavioral: Peer-Enhanced Group Exposure Therapy for Social Anxiety
- Fully enhanced (Experimental): Group exposure therapy for social anxiety and public speaking fears plus self-compassion exercises aimed at inducing a sense of common humanity, facilitated by a pair of doctoral student and undergraduate student co-facilitators who will explicitly use appropriate self-disclosure to establish the co-facilitators as individuals with lived experiences of social anxiety and public speaking fears.
  Interventions: Behavioral: Peer and Self-Compassion Enhanced Group Exposure Therapy for Social Anxiety

INTERVENTIONS:
Behavioral: Group Exposure for Social Anxiety — Group exposure therapy for social anxiety and public speaking fears.
  Arms: Exposure Only
Behavioral: Self-Compassion Enhanced Group Exposure Therapy for Social Anxiety — Group exposure therapy for social anxiety and public speaking fears plus piloted exercises from the investigators' previous studies among socially anxious undergraduates (Slivjak et al., 2022; Slivjak & Arch, in preparation), refined during the investigators' quality improvement project, that are designed to enhance compassion.
  Arms: Compassion Enhanced
Behavioral: Peer-Enhanced Group Exposure Therapy for Social Anxiety — Group exposure therapy for social anxiety and public speaking fears facilitated by a pair of doctoral student and undergraduate student co-facilitators who explicitly use appropriate self-disclosure to establish the co-facilitators as individuals with lived experiences of social anxiety and public speaking fears.
  Arms: Peer enhanced
Behavioral: Peer and Self-Compassion Enhanced Group Exposure Therapy for Social Anxiety — Group exposure therapy for social anxiety and public speaking fears plus piloted exercises from the investigators' previous studies among socially anxious undergraduates (Slivjak et al., 2022; Slivjak & Arch, in preparation), refined during the investigators' quality improvement project, that are designed to enhance compassion. These groups are facilitated by a pair of doctoral student and undergraduate student co-facilitators who explicitly use appropriate self-disclosure to establish the co-facilitators as individuals with lived experiences of social anxiety and public speaking fears.
  Arms: Fully enhanced

SUMMARY:
The purpose of the study is to investigate the effects of four versions of a workshop for social anxiety and public speaking stress. All participants are current University of Colorado Boulder undergraduate students. Participation in this research study lasts for approximately 8 weeks, and includes a pre-workshop questionnaire, 3 weekly workshop sessions (ranging from 2 to 3 hours each, including a 5-minute post-session questionnaire), a post-workshop questionnaire, and a 1-month follow-up questionnaire.

DETAILED DESCRIPTION:
The present study seeks to evaluate the feasibility, acceptability, and efficacy potential of a full factorial trial of a peer-led common humanity- and exposure-based workshop for social anxiety within a Multiphase Optimization Strategy (MOST) trial framework. The present study seeks to enroll and randomize participants (up to N = 200) by cohort to one of four conditions, reflecting a full factorial trial design. The inclusion of common humanity enhancements and the presence of a peer leader will each serve as independent variables, comprising of the following four study conditions: 1) common humanity with peer leader, 2) common humanity without peer leader, 3) peer leader without common humanity, and 4) exposure only (no common humanity and no peer leader). The investigators will assess outcomes after the workshop sessions (mid1, mid2, mid3, Post[T1]) and one-month following the conclusion of the last workshop session (T2).

The study has the following aims and hypotheses:

Aim 1: To evaluate the feasibility and acceptability of conducting a full factorial trial of a group exposure workshop for social anxiety within a MOST trial framework.

Hypothesis 1a (feasibility): At least 50% of screened, eligible participants will enroll in the study.

Hypothesis 1b (feasibility): Enrolled research participants will attend on average at least 2 out of 3 workshop sessions.

Hypothesis 1c (feasibility): Workshops will be delivered with high fidelity (80% of content checklist items covered, on average) and low contamination (20% or less inclusion of content specific to other conditions, on average) in each randomized condition.

Hypothesis 1d (acceptability): Participants will report a median satisfaction with the workshops of 4 or higher on the 1-5 Acceptability of Intervention Measure (AIM).

Hypothesis 1e (acceptability): Participation in the group workshops will be acceptable, indicated by high overall satisfaction with the workshop across conditions (mean rating of >20 on the Client Satisfaction Questionnaire-8).

Hypothesis 1f (acceptability): ≤20% of participants will report a study burden of 4 or higher on a 1-5 burden measure.

Aim 2: To evaluate the feasibility and efficacy potential of primary and secondary outcomes. Please note that the investigators do not expect to find statistically significant differences between conditions in this pilot study - only patterns of differences in the predicted directions outlined below. This pilot study will establish the foundation for a larger, definitively powered, future trial.

Hypothesis 2a (Feasibility of assessment): At least 70% of participants will complete pre, post, and follow-up surveys.

Hypothesis 2b (Efficacy potential): Compared to the exposure only condition, reliable change magnitudes (Jacobson & Truax, 1991) will be higher within the peer and compassion-enhanced conditions, with additive effects for the fully enhanced condition, on measures of 1) participant retention, 2) social anxiety, 3) depression, and 4) self-compassion.

Hypothesis 2c (Cultivating community): Compared to the exposure-only condition, reliable change magnitudes will be higher within the peer and compassion-enhanced conditions, with additive effects for the fully enhanced condition, on measures of 1) stigma and 2) sense of belonging.

Hypothesis 2d (Barriers to access and engagement): Compared to the exposure only condition, reliable change magnitudes will be higher in the peer and compassion-enhanced conditions, with additive effects for the fully enhanced condition, on measures of 1) enjoyableness, 2) likelihood to recommend, and 3) readiness and willingness to engage in therapy. Across conditions, participants will indicate a preference for peer co-facilitators over mental health providers only.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18-30
* Able to read and write fluently in English
* Current undergraduate students at CU
* Experiencing elevated social anxiety symptoms indicated by a SPIN score ≥ 19
* Experiencing moderate to high communication anxiety indicated by a PRCA- 24 score ≥ 59
* Open to receiving help for social anxiety or public speaking fears indicated by a help seeking score of ≥ 3 out of 5 (at both screening timepoints as explained below)
* Able to voluntarily consent to participation
* Able to participate fully in the study (including in the in-person group workshops and in survey completion) as assessed by screening questions and the study P

Exclusion Criteria:

* Are currently experiencing moderately severe or severe depression represented by the validated cutoff score for major depression on the PHQ-8 of greater than 14 (Kroenke et al., 2001)
* Score in the moderate-high range for suicide risk as indicated by the CSSRS (Salvi, 2019), report a suicide attempt in the past 12 months, or report current, ongoing suicidal ideation along with a past (lifetime) suicide attempt
* Are current students of the PI or clients or current students of the doctoral student co-facilitators

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Attendance rate | 3 weeks during the intervention (workshops 1, 2, and 3, 1 week apart)
  Average number of workshop sessions attended by enrolled research participants.
Enrollment rate | Pre-intervention (from screening to enrollment)
  Ratio of screened, eligible participants who enrolled in the study.
Acceptability of Intervention Measure (AIM) | 48 hours after the final intervention session and 1-month follow-up
  Workshop satisfaction rating, Range = 1 - 5, Higher scores indicate better outcome (greater acceptability)
Client Satisfaction Questionnaire-8 (CSQ-8) | 48 hours after the final intervention session and 1-month follow-up
  Satisfaction with workshops, Range = 8 - 32, Higher scores indicate better outcome (greater satisfaction)
Social Phobia Inventory (SPIN) | 48 hours after the final intervention session and 1-month follow-up
  Social anxiety symptom measure, Range = 0 - 68, Higher scores indicate worse outcome (worse social phobia)
Liebowitz Social Anxiety Scale (LSAS) | 48 hours after the final intervention session and 1-month follow-up
  Measure assessing fear/anxiety across a broad range of social and performance situations, Range = 0 - 144, Higher scores indicate worse outcome (worse social anxiety)

SECONDARY OUTCOMES:
Personal Report of Communication Apprehension (PRCA-24) | 48 hours after the final intervention session and 1-month follow-up
  Measure of trait communication and public speaking anxiety, Range = 24 - 120, Higher scores indicate worse outcome (greater communication apprehension)
Fidelity | 3 weeks during the intervention (workshops 1, 2, and 3, 1 week apart)
  Percentage of content checklist items covered during in-person workshops.
Contamination | 3 weeks during the intervention (workshops 1, 2, and 3, 1 week apart)
  Percentage of content specific to other conditions covered in each randomized condition.
Study Burden | 48 hours after the final intervention session and 1-month follow-up
  Rating of study burden.
Survey Completion | between 10 and 0 days before the first intervention session, 48 hours after the final intervention session, and 1-month follow-up
  Percentage of participants who complete pre, post, and follow-up surveys.
Participant Retention | 3 weeks during the intervention (workshops 1, 2, and 3, 1 week apart)
  Percentage of participants who completed workshops.
Patient Health Questionnaire-8 (PHQ-8) | 48 hours after the final intervention session and 1-month follow-up
  Measure of depressive symptoms, Range = 0 - 24, Higher scores indicate worse outcome (worse depression)
Self-Compassion Scale - Short (SCS) | 48 hours after the final intervention session and 1-month follow-up
  Measure of trait self-compassion and common humanity, Range = 1 - 5, Higher scores indicate better outcome (greater self-compassion)
Stigma and Self-Stigma Scale, help seeking behaviors and self-stigma subscales (SASS) | 48 hours after the final intervention session and 1-month follow-up
  Measure of stigma toward mental health problems.
  Help-seeking behaviors subscale: Range = 0 - 24, Higher scores indicate worse outcome (worse help-seeking behaviors)
  Self-stigma subscale: Range = 0 - 24, Higher scores indicate worse outcome (greater self-stigma)
Sense of Belonging Scale | 48 hours after the final intervention session and 1-month follow-up
  Measure of how connected participants feel to their group members, Range = 1-7, Higher = Higher scores indicate better outcome (greater sense of belonging)
Likelihood to Recommend | 48 hours after the final intervention session and 1-month follow-up
  Rating of how likely participants would be to recommend the workshop to others.
Enjoyableness | 48 hours after the final intervention session and 1-month follow-up
  Rating of degree to which participants found the workshop to be enjoyable.
Provider preference | between 0 and 10 days before the first intervention session, 48 hours after the final intervention session, and 1-month follow-up
  Rating of whether participants have a preference for peer co-facilitators over mental health providers only.

CONTACTS AND LOCATIONS:
Locations (1):
- Renee Crown Wellness Institute and Department of Psychology & Neuroscience, University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No